CLINICAL TRIAL: NCT04821076
Title: Influence of Low Energy Availability on Performance and Health in Trained and Recreationally Active Women
Brief Title: Influence of Low Energy Availability on Skeletal Muscle and Cardiovascular Health
Acronym: LEA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: University of Copenhagen (Other); University of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LEA
Record Dates: First submitted 2021-03-24; First posted 2021-03-29 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Diet; Deficiency; Exercise Intervention
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Intervention Model Description: Energy balance group vs. energy restriction
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Energy balance (Active Comparator)
  Interventions: Other: Diet intervention - Energy balance
- Energy restriction (Experimental)
  Interventions: Other: Diet intervention - caloric restriction
- Energy balance + exercise (Active Comparator)
  Interventions: Other: Exercise intervention; Other: Diet intervention - Energy balance
- Energy restriction + exercise (Experimental)
  Interventions: Other: Diet intervention - caloric restriction; Other: Exercise intervention

INTERVENTIONS:
Other: Diet intervention - caloric restriction — Energy restriction is set to 25 kcal / kg fat-free mass
  Arms: Energy restriction; Energy restriction + exercise
Other: Exercise intervention — Exercise will consist of supervised resistance training, interval training and moderate intensity cycling
  Arms: Energy balance + exercise; Energy restriction + exercise
Other: Diet intervention - Energy balance — Energy balance is set to 50 kcal / kg fat-free mass
  Arms: Energy balance; Energy balance + exercise

SUMMARY:
The project is designed as a randomized controlled intervention trial in which 60 young trained (n = 30) (Population A) and recreationally active (n = 30) women (Population B) with regular menstruation are divided into four groups. Population A will receive a low-calorie diet + exercise or an energy balanced diet + exercise over 10 days. Population B will receive a low-calorie diet without exercise, or an energy balanced diet over 10 days. The participants are matched in pairs based on training history and randomized. Before the diet period, the groups will undergo a 6-day control period, during which all participants must take an energy-balanced diet (± training). After the 10 days of the diet intervention period, the groups will receive an energy-balanced diet for 2 days. Before, during, and after the trial period, participants will perform performance tests. In addition, 3 muscle biopsies, 2 adipose biopsies, blood samples, urine samples will be taken during the period, as well as resting metabolic rate, electrocardiogram, flow-mediated vasodilation, and body composition over the trial period. Muscle protein synthesis rate will be measured over the period using stable isotope technique, which includes ingestion of heavy water (D2O) and collection of saliva samples daily (days 0 to 16). The primary measurement parameter is changes in muscle protein synthesis rate.

ELIGIBILITY:
Inclusion Criteria:

* age 18-30
* BMI 18.5-30
* Regular training at least 4 times a week and a maximum of 10 times a week (≥1 times strength training, ≥1 times endurance training / interval training or interval-based sports

Exclusion Criteria:

* • Irregular menstruation within the last 6 months (shorter end 24 days or longer end 35 days cycle)

  * Used hormonal contraception within the last 3 months for the trial.
  * Injuries / pain in the lower body, which prevents participation in intense strength training
  * Medication consumption that may affect protein metabolism and inflammatory parameters.
  * Diabetes
  * Smoking
  * Unstable weight / major weight loss (weight fluctuations of more than 5 kg in the last six months)
  * Do not eat animal products
  * Eating disorder
  * Pregnancy
  * Blood donor within the last month
  * Cannot read or understand Danish

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2023-06-16 (Actual)

PRIMARY OUTCOMES:
Changes in muscle protein synthesis | 10 days of diet+exercise intervention

SECONDARY OUTCOMES:
Markers of muscle protein synthesis and breakdown | before and after 10 days of diet+exercise intervention
Muscle glycogen and lipid levels | before and after 10 days of diet+exercise intervention
Sarcoplasmic reticulum function | before and after 10 days of diet+exercise intervention
Macrophage content in adipose tissue | before and after 10 days of diet+exercise intervention
Adipocyte area and cell size in adipose tissue | before and after 10 days of diet+exercise intervention
Expression of fat oxidative proteins in adipose tissue | before and after 10 days of diet+exercise intervention
Maximal isometric and dynamic muscle strength | before and after 10 days of diet+exercise intervention and 2 days of energybalance
Maximal vertical jump height | before and after 10 days of diet+exercise intervention and 2 days of energybalance
Repeated sprint ability | before and after 10 days of diet+exercise intervention and 2 days of energybalance
4-minute time trial performance | before and after 10 days of diet+exercise intervention and 2 days of energybalance
Sex hormone levels | During the course of the whole intervention period (18 days)
Cortisol Levels | During the course of the whole intervention period (18 days)
Inflammatory levels | before and after 10 days of diet+exercise intervention and 2 days of energybalance
Bone turnover levels | before and after 10 days of diet+exercise intervention and 2 days of energybalance
Electrocardiogram - Qt interval | before and after 10 days of diet+exercise intervention and 2 days of energybalance
Flow mediated vasodilation | before and after 10 days of diet+exercise intervention and 2 days of energybalance
Resting metabolic rate | before and after 10 days of diet+exercise intervention and 2 days of energybalance
Body composition | before and after 10 days of diet+exercise intervention and 2 days of energybalance

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University, Department for Public Health, Section for Sport Science, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Undecided